CLINICAL TRIAL: NCT02063438
Title: Thoracotomy Closure Technique and Postoperative Pain Study: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jules Lin, Assistant Professor; Surgical Director, Lung Transplant, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00082406
Record Dates: First submitted 2014-01-30; First posted 2014-02-14 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Hernia; Lung Cancer
Keywords: Thoracotomy; Pain; Intracostal Suture; Pericostal Suture
MeSH Terms: conditions — Hernia; Lung Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pericostal Suture Technique (Active Comparator): A #2 Vicryl suture is placed along the superior aspect of the rib above the specific thoracic interspace. This suture is then passed below the inferior rib along the superior aspect of the next rib below. These sutures are then tied to approximate the ribs leaving enough room for the tip of a finger.
  Interventions: Procedure: Pericostal suture technique
- Intracostal Suture Technique (Active Comparator): A handheld drill is used to drill holes in the rib below the specific thoracic interspace. A #2 Vicryl suture is passed through each of the holes and then passed along the superior aspect of the rib above the specific thoracic interspace. These sutures are then tied to approximate the ribs leaving enough room for the tip of a finger.
  Interventions: Procedure: Intracostal suture technique

INTERVENTIONS:
Procedure: Pericostal suture technique
  Arms: Pericostal Suture Technique
Procedure: Intracostal suture technique
  Arms: Intracostal Suture Technique

SUMMARY:
The purpose of this study is to examine pain associated with thoracotomy (incision made during surgery to obtain access to your thoracic cavity) and how the closure technique may influence postoperative pain. Two types of routinely selected thoracotomy closure techniques will be examined; pericostal and intracostal sutures. The investigators hypothesize that intracostal sutures will result in less postoperative and chronic pain as a result of less compression of the intercostal nerve.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective procedure that will include a thoracotomy.
* All patients will undergo epidural catheter placement.

Exclusion Criteria:

* Previous thoracotomy on the operative side.
* Previous history of chronic chest pain.
* Previous history of thoracic trauma on the operative side.
* Less than 18 years of age
* Inability to provide informed consent or to complete testing or data collection
* Need for a chest wall resection
* Patients requiring other incisions in addition to a thoracotomy (i.e., Laparotomy, sternotomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Severity of postoperative pain in the perioperative period. | 2 weeks following surgery
Intensity and incidence of chronic post-thoracotomy pain | 6 months follwong surgery

SECONDARY OUTCOMES:
Complication rates between subjects undergoing pericostal versus intracostal thoracotomy closure technique | 6 months following surgery
Length of hospital stay and associated hospital costs between subjects undergoing pericostal versus intracostal thoracotomy closure technique | 6 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jules Lin, MD, Principal Investigator — UM Department of Surgery, Section of Thoracic Surgery
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Allama AM. Intercostal muscle flap for decreasing pain after thoracotomy: a prospective randomized trial. Ann Thorac Surg. 2010 Jan;89(1):195-9. doi: 10.1016/j.athoracsur.2009.07.094. PMID 20103234
- [Background] Sakakura N, Usami N, Taniguchi T, Kawaguchi K, Okagawa T, Yokoyama M, Yokoi K. Assessment of long-term postoperative pain in open thoracotomy patients: pain reduction by the edge closure technique. Ann Thorac Surg. 2010 Apr;89(4):1064-70. doi: 10.1016/j.athoracsur.2010.01.015. PMID 20338308
- [Result] Cerfolio RJ, Price TN, Bryant AS, Sale Bass C, Bartolucci AA. Intracostal sutures decrease the pain of thoracotomy. Ann Thorac Surg. 2003 Aug;76(2):407-11; discussion 411-2. doi: 10.1016/s0003-4975(03)00447-8. PMID 12902074
- [Result] Cerfolio RJ, Bryant AS, Maniscalco LM. A nondivided intercostal muscle flap further reduces pain of thoracotomy: a prospective randomized trial. Ann Thorac Surg. 2008 Jun;85(6):1901-6; discussion 1906-7. doi: 10.1016/j.athoracsur.2008.01.041. PMID 18498792
- [Result] Cerfolio RJ, Bryant AS, Patel B, Bartolucci AA. Intercostal muscle flap reduces the pain of thoracotomy: a prospective randomized trial. J Thorac Cardiovasc Surg. 2005 Oct;130(4):987-93. doi: 10.1016/j.jtcvs.2005.05.052. PMID 16214509
- [Result] Bayram AS, Ozcan M, Kaya FN, Gebitekin C. Rib approximation without intercostal nerve compression reduces post-thoracotomy pain: a prospective randomized study. Eur J Cardiothorac Surg. 2011 Apr;39(4):570-4. doi: 10.1016/j.ejcts.2010.08.003. Epub 2010 Sep 15. PMID 20833556
- [Result] Wu N, Yan S, Wang X, Lv C, Wang J, Zheng Q, Feng Y, Yang Y. A prospective, single-blind randomised study on the effect of intercostal nerve protection on early post-thoracotomy pain relief. Eur J Cardiothorac Surg. 2010 Apr;37(4):840-5. doi: 10.1016/j.ejcts.2009.11.004. Epub 2009 Dec 1. PMID 19954996
- [Result] Gordon DB, Polomano RC, Pellino TA, Turk DC, McCracken LM, Sherwood G, Paice JA, Wallace MS, Strassels SA, Farrar JT. Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) for quality improvement of pain management in hospitalized adults: preliminary psychometric evaluation. J Pain. 2010 Nov;11(11):1172-86. doi: 10.1016/j.jpain.2010.02.012. Epub 2010 Apr 18. PMID 20400379